CLINICAL TRIAL: NCT03971461
Title: A Single Arm, Open-label, Multicenter Phase II Study of 177Lu-DOTATATE Radionuclide in Adults With Progressive or High-risk Meningioma
Brief Title: Phase II Study of 177Lu-DOTATATE Radionuclide in Adults With Progressive or High-risk Meningioma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-00719
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Intervention Model Description: Open-label, single arm, multicenter, two-stage phase 2 clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lutathera (Experimental)
  Interventions: Drug: Lutathera

INTERVENTIONS:
Drug: Lutathera — administered intravenously every 8 weeks for a total of 4 doses
  Other Names: 177Lu-DOTATATE

SUMMARY:
This single arm, open-label study will evaluate the efficacy of Lutathera (177Lu-DOTATATE) administered intravenously every 8 weeks for a total of 4 doses in patients with progressive WHO I-III or residual high-risk Ga-DOTATATE PET-MRI positive meningioma. Ga-DOTATATE PET-MRI scans will be obtained prior to initiation of Lutathera treatment and 6 months after the initiation of Lutathera treatment. The latter will be performed within the 14 days prior to the last dose of Lutathera treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years.
2. Karnofsky Performance Status ≥ 60.
3. Histologically confirmed diagnosis WHO grade I-III meningioma:

   a. For grade I meningioma, subjects must have: i. Progressive disease after at least surgical resection and radiotherapy, as defined as an increase in size of the measurable primary lesion (bidirectional area) on imaging by 25% or more between scans separated by no more than 12 months.

   or ii. Progressive residual tumor after maximal safe resection, be located at or near critical organs at-risk and considered to be high-risk for radiation injury by the treating investigator. Prior external beam radiotherapy is not required for these subjects.

   b. For Grade II or III meningioma, subjects must have either: i. Progressive disease after at least surgical resection and radiotherapy, as defined as an increase in size of the measurable primary lesion (bi-directional area) on imaging by 25% or more between scans separated by no more than 12 months or ii. Residual measurable disease after surgery without requirement of progression.
4. Positive 68Ga-DOTATATE uptake on PET-MRI.

   1. Positive uptake is defined as uptake higher than the background and SUV ratios adjusted to the liver and spleen uptake (adopted from Krenning score).
   2. 68Ga-DOTATATE uptake in target lesions should be Krenning score ≥ 2.
5. Presence of measurable disease defined as at least one lesion measuring ≥10 mm in at least one dimension by contrast-enhanced MRI performed within 30 days prior to study registration.
6. Multifocal disease is allowed but is limited to ≤ 3 measurable intracranial mass lesions on the most recent post-contrast MRI.
7. Any neurological symptoms must be stable for at least 28 days prior to enrollment and patients should not require steroids to control neurological symptoms.
8. There is no limit on the number of prior surgeries, radiation therapy, radiosurgery treatments or systemically administered therapeutic agents.
9. For patients treated with external beam radiation, interstitial brachytherapy or radiosurgery, an interval ≥24 weeks must have elapsed from completion from these therapies to registration unless there is histopathologic confirmation of recurrent tumor or there is new enhancing tumor outside the radiation field (beyond the high dose region or the 80% isodose line).
10. An interval of ≥28 days (or 5 half-lives, whichever is shorter) from prior cytotoxic chemotherapy (6 weeks from nitrosoureas), biologic agent, investigational agent or any other systemic agent prescribed for the purpose of treating meningioma.
11. An interval of ≥28 days from craniotomy and ≥7 days from stereotactic biopsy.
12. Availability of a paraffin-embedded archival tumor block from most recent tumor resection sufficient to generate at minimum 8 unstained slides but preferably up to 25 unstained slides; or, if a paraffin tumor block is unavailable, at minimum 8 unstained slides but preferably up to 25 unstained slides.

    a. Positive SSTR2 expression in the most recent tumor specimen must be confirmed by central pathology review.
13. Patients must be willing and able to undergo regular MRI scans of the brain.
14. Patients must have recovered to CTCAE grade ≤1 or pretreatment baseline from clinically significant adverse events related to prior therapy (exclusions include alopecia, laboratory values listed per inclusion criteria, lymphopenia, sensory neuropathy ≤ grade 2, or other ≤ grade 2 not constituting a safety risk based on the investigator's judgment).
15. Adequate organ and bone marrow function as defined below (within 21 days of treatment initiation):

    1. White blood cell (WBC) ≥ 2,000/mm3
    2. Absolute neutrophil count (ANC) ≥ 1,000/mm3
    3. Platelet count ≥ 75,000/mm3
    4. Hemoglobin ≥ 8 gm/dL
    5. AST(SGOT)/ALT(SGPT) ≤ 3 x laboratory upper limit of normal (ULN)
    6. Creatinine clearance (measured or calculated) ≥ 50 mL/min OR creatinine levels > 150 μMol/L (1.7 mg/dL)
    7. Total serum bilirubin ≤ 3 X ULN (except participants with Gilbert's Syndrome, who can have a total bilirubin ≤ 5 X ULN)
    8. Serum albumin level of more than 3.0 g/dL, unless the prothrombin time value was within the normal range
16. Women of childbearing potential (WOCBP) and men able to father a child must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in the study, she must inform her treating physician immediately.
17. Able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria

1. Patients with a clinical diagnosis of NF2 (either by NIH or Manchester criteria) or with a molecular diagnosis of NF2.
2. Patients with radiation-associated meningiomas.
3. Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm. This includes treatment with Somatostatin LAR within 4 weeks prior to treatment, or any patient receiving treatment with short-acting Octreotide that cannot be interrupted for greater than 24 hours before treatment.
4. Peptide receptor radionuclide therapy at any time prior to registration.
5. Known hypersensitivity to somatostatin analogues or any component of the 68Ga- DOTATATE or 177Lu-DOTATATE formulations.
6. Known additional malignancy that is progressing or requires active treatment within 2 years of start of study drug. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and in situ cervical cancer that has undergone potentially curative therapy.
7. Current or planned participation in another study of an investigational agent or investigational device.
8. Active infection requiring intravenous therapy with antibiotics.
9. Uncontrolled intercurrent illness including, but not limited to, clinically significant (i.e. active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), congestive heart failure (≥ NYHA class II), unstable angina pectoris, or serious cardiac arrhythmia requiring medication.
10. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
11. Active Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test is positive).
12. Other severe acute or chronic medical or psychiatric conditions (within the past year) including recent or active suicidal ideation or behavior, or laboratory abnormalities that may increase the risk associated with study participation or treatment on study or may interfere with the interpretation of study results.
13. Pregnant and/or breastfeeding patients. Women of childbearing potential (WOCBP) must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival at 6 months (PFS-6) | 6 Months
  proportion of subjects who achieve a complete response (CR), partial response (PR), or stable disease (SD) at 6 months from start of Lutathera treatment. Radiographic treatment response will be assessed by measuring the bidirectional tumor diameters on contrast-enhanced MRI in patients who received at least one dose of Lutathera compared to baseline measurements at time of study enrollment

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 12 months
  defined as the best response [Complete Response (CR) + Partial Response (PR) + stable disease (SD)] recorded from the start of the study until the end of study in patients who received at least one dose of Lutathera.
Overall Survival at 12 months (OS-12) | 12 months
  proportion of subjects who are alive at 12 months from start of Lutathera treatment. Survival data will be captured by clinical follow-up every 8 weeks during treatment with Lutathera and by follow-up phone calls every 12 weeks for up to 2 years after completion of treatment with Lutathera.
Progression Free Survival (PFS) | 2 Years Post Treatment
  defined as the number of days from the treatment start date to the date of documented disease progression or death due to any cause.
Overall Survival (OS) | 2 Years Post Treatment
  defined as the number of days from the treatment start date to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Sulman, MD, Principal Investigator — New York Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - Cleveland Clinic, Cleveland, Ohio